CLINICAL TRIAL: NCT03953144
Title: Synapse 3D With Intravascular Indocyanine Green Fluorescence Mapping for Targeted Pulmonary Segmental Resection Trial: A Phase I Safety and Feasibility Trial
Brief Title: Synapse 3D With Intravascular Indocyanine Green
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Wael Hanna, Director, Research Program, Boris Family Centre for Robotic Surgery, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VISION10042019
Record Dates: First submitted 2019-04-30; First posted 2019-05-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer; Primary Neoplasm
Keywords: Segmentectomy; Lung Cancer; Robotic Surgery; 3D Modelling; CT Imaging; Near-Infrared Fluorescence; IC-GREEN; Surgical Planning; Indocyanine Green; Early-Stage Lung Cancer; Surgical Mapping; Lung Preservation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: This study is a single centre, prospective clinical trial evaluating the safety and feasibility of adding 3D anatomical reconstructions and real-time intraoperative planning using Synapse 3D software added to NIF-guided targeted segmental resection. It is anticipated that 32 participants will be enrolled within a 1-year period. Enrollment will take place at St. Joseph's Healthcare Hamilton. All patients enrolled will be evaluated until their first scheduled follow-up appointment (within 30 days post-surgery).
Masking Description: Open Label, single-arm feasibility trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Synapse 3D Lung Modelling + IC-GREEN Segmentectomy (Experimental): Patients within this arm will undergo a high-resolution CT scan of the chest, which is required by Synapse 3D to create accurate 3D virtual model reconstructions. At the start of the operation, the 3D virtual model of the segmental pulmonary anatomy will be displayed on the da Vinci Robotic platform for operative planning. The model will be used as a guide to determine which vessels are involved in the segment and need to be removed. The surgeon will ligate the pulmonary vein and pulmonary artery of the broncho-pulmonary segment with the lung cancer nodule, isolating it from any blood supply, and mark the proposed segmental planes based on the 3D model. ICG will be prepared as a sterile solution (2.5 mg/10mL) for injection. After vascular ligation, an 8 mL bolus of ICG solution will be injected into the peripheral vein catheter, followed by a 10 mL saline solution bolus
  Interventions: Device: Synapse 3D Lung Modelling; Drug: IC-Green (ICG)

INTERVENTIONS:
Device: Synapse 3D Lung Modelling — The 3D virtual models provided by Synapse 3D will be made by experts in medical image analysis using the high-resolution CT scans. Patients will have 3D virtual reconstructions of their pulmonary anatomy with the target lesion created pre-operatively.
Drug: IC-Green (ICG) — ICG will be prepared as a sterile solution (2.5 mg/10mL) for injection. After vascular ligation, a 6 to 8mL bolus of ICG solution will be injected into the peripheral vein catheter, followed by a 10mL saline solution bolus. The Firefly camera will then be used for the NIF imaging. It is expected that the entire lung, except the segment which was previously isolated from blood supply, will fluoresce within 30-40 seconds, exhibiting a green hue. The surgeon will perform the pulmonary resection and the resected 'dark' lung segment will be immediately evaluated by a pathologist, depending on the pathologist findings the operation may be concluded or the patient will receive a pulmonary lobectomy.
  Other Names: Indocyanine Green

SUMMARY:
With the advent of CT screening for lung cancer, an increasing number of NSCLCs are being detected at very early stages, and the demand for pulmonary segmentectomy is rising rapidly. As such, there is a need to develop new surgical techniques to facilitate minimally invasive pulmonary segmentectomy, as segmentectomy may provide a number of significant advantages over lobectomy for patients presenting with early-stage lung cancer, or for patients unable to undergo a full lobectomy due to existing comorbidities. This study will provide the first case series using preoperative 3D anatomical planning (Synapse 3D) added to ICG and NIF-guided robotic segmentectomy to date and will be the first reported use of Synapse 3D-guided targeted pulmonary segmental resection in Canada. As lung cancer is the most frequently fatal cancer in North America, many thousands of patients will be able to benefit from this operation every year.

DETAILED DESCRIPTION:
Lungs are made up of individual lobes. When a lung cancer tumour is found in one of these lobes, the surgeon often performs a Lobectomy. A Lobectomy is the surgery most commonly done to treat early-stage lung cancer and requires removal of an entire lobe of the lung, which removes a large amount of lung tissue

For patients with small tumours saving as much healthy lung tissue as possible is important. Each lobe of the lung has smaller sections called segments. When a lung cancer is in one of these segments, it is possible to remove that segment, without removing the entire lobe. This surgery is called a Segmentectomy. Compared to a lobectomy, a segmentectomy saves a larger amount of healthy lung tissue. Research shows that a segmentectomy can result in less blood loss, shorter operation time, less days of having a chest tube, and a shorter hospital stay, compared to a lobectomy.

With the advances in screening technology for lung cancer tumours, an increasing amount of very small lung cancer tumours are being found, and the demand for segmentectomy is increasing. A segmentectomy is a hard surgery to perform robotically because it is difficult to view the tissue lines that separate each segment within the lobe. As a result, it is difficult for the surgeon to see exactly which pieces of tissue should be removed in order to safely complete the segmentectomy. Because of these challenges, many patients having robotic surgery will have a lobectomy, even if a full lobectomy is not needed.

In response to these challenges, our surgical group has developed the technique of using Near-Infrared Fluorescence (NIF) mapping with intravascular indocyanine green (ICG) dye injection. With the aid of an infrared camera the surgeon is able to see the segment within a lobe of lung after injection of the ICG dye, allowing for a more accurate segmentectomy. We recently reported a 60% success rate of segmental resections with the use of ICG and NIF-guided surgical resection. However, a limitation to this technique is that the segmental anatomy can only be seen during the operation and only after cutting the blood vessels.

The introduction of 3D reconstruction and virtual modeling provides a new way to locate lesions accurately within a segment and plan the appropriate operation before the actual surgery occurs. Synapse 3D (Mississauga, Canada) is a 3D modelling technology that is capable of producing a detailed 3D virtual model of a patient's lung based on Computed Tomography (CT) scans. It has been shown to be safe and feasible in performing segmental pulmonary resections on a robotic platform. In this study, we propose a new operation that uses 3D anatomical planning before the surgery (Synapse 3D) and real-time NIF-mapping at the time of surgery using ICG dye, which we believe will greatly increase the likelihood of a successful segmentectomy. If this new operation is successful, it will help patients save more of their healthy lung tissue when they are undergoing surgery for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Tumour size <3 cm
* Clinical Stage 1 Non-Small Cell Lung Cancer (NSCLC)
* CT-imaging confirming that the tumour is confined to one broncho-pulmonary segment, rendering the patient a candidate for segmental resection.

Exclusion Criteria:

* Hypersensitivity or allergy to ICG, sodium iodide, or iodine
* Women who are currently pregnant or breastfeeding; or women of childbearing potential who are not currently taking adequate birth control.
* Patients with clinical evidence of N1 or N2 disease on preoperative imaging
* Pulmonary Function tests demonstrating Forced Expiratory Volume in 1s (FEV1) or diffusion capacity of the lung for carbon monoxide (DLCO) less than or equal to 30% of predicted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Segmental Resection Conversion Rate | 1 year
  Rate of conversions to lobectomy will be measured by collecting the proportion of conversions to lobectomy.
Number of Participants with Post Operative Complications | 1 year
  Post operative complications will be reported and measured using the Ottawa Thoracic Morbidity and Mortality Classification of (a) Adverse reactions to ICG dye at the time of surgery and (b) Perioperative complications through study completion.

SECONDARY OUTCOMES:
Anatomical Accuracy of the 3D Lung Model | 1 year
  Anatomical accuracy will be evaluated using the criteria listed in points a-c. A score of 3/3 on these items will indicate success of anatomical accuracy
  1. Ex-vivo localization of lesions;
  2. Ex-vivo confirmation of tumor-free margins around lesion;
  3. Ex-vivo confirmation of adequate anatomical inter-segmental.
Surgeon Confidence | 1 year
  A pre-operative CT scan based, a pre-operative 3D reconstruction based and post segmental resection surgeon confidence score will be obtained on a scale of 1-5:
  1 - not at all confident, 2 - somewhat confident, 3 - confident, 4 - very confident, 5 - extremely confident.
Operation Time | 1 year
  Length of time of the operation will be measured by collecting the time the patient entered the operating room until the time the patient left the operating room.
Conversion to Thoracotomy | 1 year
  Rate of conversion to thoracotomy will be measured by collecting the proportion of conversions to thoracotomy. Descriptive analysis of reasons for conversion will also be collected.
Chest Tube Duration | 1 year
  Duration the patient had chest tubes in situ will be measured by collecting the date of surgery and the date the chest tube was removed.
Length of Stay | 1 year
  Duration of hospital length of stay will be measured by collecting the data of admission and the date of discharge.
Estimated Blood Loss | 1 year
  Estimated blood loss will be measured at the time of operation by OR staff.

CONTACTS AND LOCATIONS:
Overall Officials: Waël C Hanna, MDCM, MBA, FRCSC, Principal Investigator — St. Joseph's Healthcare Hamilton / McMaster University
Locations (1):
- St. Josephs Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Landreneau RJ, Sugarbaker DJ, Mack MJ, Hazelrigg SR, Luketich JD, Fetterman L, Liptay MJ, Bartley S, Boley TM, Keenan RJ, Ferson PF, Weyant RJ, Naunheim KS. Wedge resection versus lobectomy for stage I (T1 N0 M0) non-small-cell lung cancer. J Thorac Cardiovasc Surg. 1997 Apr;113(4):691-8; discussion 698-700. doi: 10.1016/S0022-5223(97)70226-5. PMID 9104978
- [Background] Zhao X, Qian L, Luo Q, Huang J. Segmentectomy as a safe and equally effective surgical option under complete video-assisted thoracic surgery for patients of stage I non-small cell lung cancer. J Cardiothorac Surg. 2013 Apr 29;8:116. doi: 10.1186/1749-8090-8-116. PMID 23628209
- [Background] Bedetti B, Bertolaccini L, Rocco R, Schmidt J, Solli P, Scarci M. Segmentectomy versus lobectomy for stage I non-small cell lung cancer: a systematic review and meta-analysis. J Thorac Dis. 2017 Jun;9(6):1615-1623. doi: 10.21037/jtd.2017.05.79. PMID 28740676
- [Background] Gossot D, Seguin-Givelet A. Anatomical variations and pitfalls to know during thoracoscopic segmentectomies. J Thorac Dis. 2018 Apr;10(Suppl 10):S1134-S1144. doi: 10.21037/jtd.2017.11.87. PMID 29785286
- [Background] Mehta M, Patel YS, Yasufuku K, Waddell TK, Shargall Y, Fahim C, Hanna WC. Near-infrared mapping with indocyanine green is associated with an increase in oncological margin length in minimally invasive segmentectomy. J Thorac Cardiovasc Surg. 2019 May;157(5):2029-2035. doi: 10.1016/j.jtcvs.2018.12.099. Epub 2019 Jan 21. PMID 30803778
- [Background] Fukuhara K, Akashi A, Nakane S, Tomita E. Preoperative assessment of the pulmonary artery by three-dimensional computed tomography before video-assisted thoracic surgery lobectomy. Eur J Cardiothorac Surg. 2008 Oct;34(4):875-7. doi: 10.1016/j.ejcts.2008.07.014. Epub 2008 Aug 15. PMID 18703345
- [Background] Baste JM, Soldea V, Lachkar S, Rinieri P, Sarsam M, Bottet B, Peillon C. Development of a precision multimodal surgical navigation system for lung robotic segmentectomy. J Thorac Dis. 2018 Apr;10(Suppl 10):S1195-S1204. doi: 10.21037/jtd.2018.01.32. PMID 29785294
- [Background] Ivanovic J, Al-Hussaini A, Al-Shehab D, Threader J, Villeneuve PJ, Ramsay T, Maziak DE, Gilbert S, Shamji FM, Sundaresan RS, Seely AJ. Evaluating the reliability and reproducibility of the Ottawa Thoracic Morbidity and Mortality classification system. Ann Thorac Surg. 2011 Feb;91(2):387-93. doi: 10.1016/j.athoracsur.2010.10.035. PMID 21256276
- [Background] Pardolesi A, Veronesi G, Solli P, Spaggiari L. Use of indocyanine green to facilitate intersegmental plane identification during robotic anatomic segmentectomy. J Thorac Cardiovasc Surg. 2014 Aug;148(2):737-8. doi: 10.1016/j.jtcvs.2014.03.001. Epub 2014 Mar 5. No abstract available. PMID 24680390